CLINICAL TRIAL: NCT02097043
Title: A Block-randomized, Double-blind, Placebo-controlled, Single-dose, Phase I Clinical Study to Investigate the Pharmacokinetics and Safety/Tolerability of DA-7218 in Healthy Male Volunteers
Brief Title: Phase I Clinical Study to Investigate the Pharmacokinetics and Safety/Tolerability of DA-7218 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: DA7218_PK_I
Record Dates: First submitted 2014-03-24; First posted 2014-03-26 (Estimated); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: Healthy
MeSH Terms: interventions — tedizolid phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (6):
- [Group 1] DA-7218 (Experimental): 200mg, By mouth or orally (PO) & intravenous(IV) administration
  Interventions: Drug: DA-7218
- [Group 1] Placebo (Placebo Comparator): Placebo, By mouth or orally (PO) & intravenous(IV) administration
  Interventions: Drug: Placebo
- [Group 2] DA-7218 (Experimental): 400mg, By mouth or orally (PO) administration
  Interventions: Drug: DA-7218
- [Group 2] Placebo (Placebo Comparator): Placebo, By mouth or orally (PO) administration
  Interventions: Drug: Placebo
- [Group 3] DA-7218 (Experimental): 600mg, By mouth or orally (PO) administration
  Interventions: Drug: DA-7218
- [Group 3] Placebo (Placebo Comparator): Placebo, By mouth or orally (PO) administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DA-7218
  Arms: [Group 1] DA-7218; [Group 2] DA-7218; [Group 3] DA-7218
Drug: Placebo
  Arms: [Group 1] Placebo; [Group 2] Placebo; [Group 3] Placebo

SUMMARY:
This study is a phase I clinical trial for evaluating the pharmacokinetics and safety/tolerability of DA-7218 in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male Korean 19-45 years
* Body weight:55-90kg, BMI:18.0-27.0

Exclusion Criteria:

* Present condition or history of any clinically significant disease
* Clinical evidence or history of GI disease or history of GI surgery
* History of hypersensitivities, including drug allergies
* AST (SGOT) or ALT (SGPT) > 1.5 times the upper normal limit
* Systolic blood pressure : <100 mmHg or >160 mmHg
* Diastolic blood pressure : <60 mmHg or >100 mmHg
* Drug abuse within 2 months, or a positive reaction to an abusive drug or cotinine
* Taken any ETC or herbal supplement within 2 weeks or any OTC or vitamin supplement within 1 week
* Participation in and administration of IP of another clinical trial within 2 months
* Donation of whole blood within 2 months, or blood components within 1 month, or receipt of blood transfusion within 1 month
* Consumption of more than 21 units of alcohol/week or inability to abstain from drinking during the study period
* Smoking within 3 months
* Taking caffeine- or grapefruit-containing products within 3 days
* Plan to be pregnant, or not to use an appropriate method of contraception

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2014-05; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
AUClast | 72 hours
  Area under the concentration-time curve from time zero to the last quantifiable concentration by linear trapezoidal method
Cmax | 72 hours

SECONDARY OUTCOMES:
tmax, AUCinf, t1/2, CL/F, Vz/F (F; calculated in group 1) | 72 hours

OTHER OUTCOMES:
Adverse events (subjective or objective symptoms) | 14 days(group 1), 7 days(group 2,3)
Vital signs | 14 days(group 1), 7 days(group 2,3)
Physical examination | 14 days(group 1), 7 days(group 2,3)
12-lead ECG | 14 days(group 1), 7 days(group 2,3)
Clinical laboratory tests | 14 days(group 1), 7 days(group 2,3)

CONTACTS AND LOCATIONS:
Overall Officials: Kyung Sang Yu, M.D., Ph.D., Principal Investigator — Seoul National University College of Medicine / Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Kim Y, Kim A, Lee S, Choi SH, Lee DY, Song JS, Lee H, Jang IJ, Yu KS. Pharmacokinetics, Safety, and Tolerability of Tedizolid Phosphate After Single-dose Administration in Healthy Korean Male Subjects. Clin Ther. 2017 Sep;39(9):1849-1857. doi: 10.1016/j.clinthera.2017.08.002. Epub 2017 Aug 31. PMID 28865799